CLINICAL TRIAL: NCT07003269
Title: An Observational Study on the Promotion of Platelet Recovery by Hetrombopag During Haploidentical Hematopoietic Stem Cell Transplantation
Brief Title: Observational Study: Hetrombopag for Platelet Recovery in Haploidentical HSCT
Status: Enrolling by invitation | Type: Observational
Sponsor: Haikou Affiliated Hospital of Central South University Xiangya School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: SC20240561
Record Dates: First submitted 2025-05-15; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Thalassemia in Children
Keywords: Thalassemia; HSCT; Hetrombopag
MeSH Terms: conditions — Thalassemia | interventions — hetrombopag

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental group: In allogeneic hematopoietic stem cell transplantation, hetrombopag is initiated at 3 µg/kg subcutaneously on day +6 post-transplant. The dose is increased by 2 µg/kg weekly up to a maximum of 10 µg/kg. Treatment is discontinued when platelet counts rise to 100×10⁹/L. If platelet counts remain ≤20×10⁹/L on day +20, hetrombopag is combined with eltrombopag 25 mg orally once daily. Fresh apheresis platelet suspensions (1 therapeutic dose, containing >2.5×10¹¹ platelets) are administered when platelet counts are ≤20×10⁹/L or when counts are between 21-50×10⁹/L with active bleeding. If engraftment has not occurred by day +28 post-transplant, re-transplantation is required, and hetrombopag is considered ineffective.
  Interventions: Drug: Hetrombopag

INTERVENTIONS:
Drug: Hetrombopag — In allogeneic hematopoietic stem cell transplantation, hetrombopag is initiated at 3 µg/kg subcutaneously on day +6 post-transplant. The dose is increased by 2 µg/kg weekly up to a maximum of 10 µg/kg. Treatment is discontinued when platelet counts rise to 100×10⁹/L. If platelet counts remain ≤20×10⁹/L on day +20, hetrombopag is combined with eltrombopag 25 mg orally once daily. Fresh apheresis platelet suspensions (1 therapeutic dose, containing >2.5×10¹¹ platelets) are administered when platelet counts are ≤20×10⁹/L or when counts are between 21-50×10⁹/L with active bleeding. If engraftment has not occurred by day +28 post-transplant, re-transplantation is required, and hetrombopag is considered ineffective.
  Other Names: Hetrombopag Olamine

SUMMARY:
The objective of this observational study is to investigate the long-term effects of Hetrombopag in promoting platelet engraftment during haploidentical hematopoietic stem cell transplantation (HSCT) in children with thalassemia, with a specific focus on a 28-day time window post-transplantation. The core question to be addressed is: Is Hetrombopag safe and effective for platelet engraftment in children with thalassemia undergoing haploidentical HSCT within a 28-day post-transplant period? Subjects who received Hetrombopag as part of routine care for haploidentical HSCT in children with thalassemia will be required to complete a 28-day online survey on platelet engraftment outcomes.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) remains a critical and often the sole curative modality for diverse hematological malignancies and disorders. Post-transplant thrombocytopenia (platelet count <20×10⁹/L) significantly compromises long-term patient survival, with an incidence of 5-20% in allo-HSCT recipients, thereby escalating treatment morbidity and costs. Current research on platelet engraftment promotion in pediatric thalassemia patients undergoing allo-HSCT is limited. Repeated platelet transfusions are associated with substantial complications, including transfusion reactions, platelet alloimmunization, and transfusion-transmitted viral infections. Eltrombopag, a thrombopoietin receptor agonist (TPO-RA), carries a black-box warning for hepatotoxicity, with a real-world incidence of 11.8%. Transplant recipients frequently experience diarrhea, which impairs the absorption of oral thrombopoietic agents, while daily subcutaneous injections exacerbate pediatric patient discomfort and reduce treatment adherence. In contrast, long-acting TPO-RAs administered once post-transplant have demonstrated favorable tolerability and promising efficacy in thalassemia transplant pediatric populations. To date, clinical data on Hetrombopag use for platelet recovery in haploidentical HSCT for pediatric thalassemia are lacking. Therefore, this observational study aims to evaluate the efficacy and safety of Hetrombopag in facilitating platelet engraftment during haploidentical HSCT in children with thalassemia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with severe thalassemia via thalassemia gene testing, transfusion history, and complete blood count (CBC).
* Pediatric patients aged 2-17 years.
* Consented to haploidentical transplantation and evaluated by the transplant team as having no transplant contraindications.

Exclusion Criteria:

* Presence of a fully matched donor with refusal of haploidentical transplantation.
* Donor or recipient with transaminase levels >2× the upper limit of normal (ULN).
* Positive hepatitis B DNA test result.
* Active infection at the time of enrollment.
* Donor-specific antibodies (DSA) >5,000 and unable to decrease below 3,000 after antibody therapy.
* Presence of transplant contraindications as assessed by the transplant team.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The Department of Hematology of Haikou People's Hospital accepts children with severe thalassemia aged 2 - 17 years old for haploidentical hematopoietic stem cell transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Platelet recovery time | From enrollment to 28 days after transplantation
  The time at nodes such as platelet >20×10^9/L, 50×10^9/L and 100×10^9/L
Platelet transfusion volume | From enrollment to 28 days after transplantation
  Required dosage of platelet suspension

SECONDARY OUTCOMES:
The rate of adverse drug reactions | From enrollment to 28 days after transplantation
  The rate of adverse drug reactions occurring during the follow-up period
Bleeding incidence rate | From enrollment to 28 days after transplantation
  The incidence rate of bleeding during the follow-up period
Thrombosis incidence rate | From enrollment to 28 days after transplantation
  The incidence rate of thrombosis during the follow-up period
Survival rate | From enrollment to 28 days after transplantation
Relapse-free survival rate | From enrollment to 28 days after transplantation
Transplant-related mortality rate | From enrollment to 28 days after transplantation
Major transplant-related complications | From enrollment to 28 days after transplantation
Cause of death | From enrollment to 28 days after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyang Yang, MD, Principal Investigator — Department of Hematology, Haikou People's Hospital
Locations (1):
- Haikou Affiliated Hospital of Central South University Xiangya School of Medicine, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: No
The IPD encompasses highly sensitive and confidential data that was collected through significant investment of our resources, both in terms of time and funding. This data is integral to our ongoing research initiatives, which are at a crucial stage of development. Premature sharing could disrupt our research timelines and strategic plans. Additionally, we have not yet established comprehensive safeguards to ensure that the data will be used appropriately by external researchers. Without proper protocols in place, there is a risk of misuse or misinterpretation of the data, which could lead to inaccurate research outcomes and potential reputational damage to our institution. For these reasons, we have decided not to share the IPD at this time.